CLINICAL TRIAL: NCT03229369
Title: Association of Anterolateral Ligament and Anterior Cruciate Ligament Reconstruction Lead to Superior Outcomes and Lower Failure Rates in High-risk Population?: a Randomized Controlled Trial.
Brief Title: Association of ALL and ACL Reconstruction Versus Isolated ACL Reconstruction in High-risk Population: a RCT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fernando Cury Rezende, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anterolateral ligament trial
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Anterior Cruciate Ligament Rupture; Ligament Knee Injury
Keywords: ACL; ALL; Ligament injury; Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Surgeons and participants of the study will not be blinded due to the intrinsic characteristics of the intervention trials, in which it is impossible to blind surgeons and avoid acknowledgement of the participants of which procedure they were assigned. However, outcome evaluation will be performed by an individual who will not have acknowledgement of which group the patient was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated ACL (Active Comparator): Standard Anterior Cruciate Ligament Reconstruction only
  Interventions: Procedure: Isolated anatomic ACL reconstruction
- Combined ACL and ALL (Experimental): Anterior Cruciate Ligament Reconstruction associated with Anterolateral Ligament Reconstruction
  Interventions: Procedure: Combined Anterior Cruciate Ligament and Anterolateral Ligament reconstruction

INTERVENTIONS:
Procedure: Isolated anatomic ACL reconstruction — Hamstrings free grafts using a two-incision intra-articular Anterior Cruciate ligament (ACL) reconstruction technique. Both ST and gracilis will be prepared with doubled strands, a standard quadrupled graft. The femoral tunnel will be performed in outside-in manner. The tibial tunnel will be drilled in the center of the ACL tibial footprint, sparing the ACL tibial stump, when possible. ACL graft will be first fixed in the femur and then in the tibia, both with an interference screw at 30 degrees of knee flexion.
  Arms: Isolated ACL
Procedure: Combined Anterior Cruciate Ligament and Anterolateral Ligament reconstruction — Hamstrings free grafts using a two-incision ACL reconstruction with the addition of a gracilis prolongation for ALL reconstruction. ACL graft will exhibit a quadruple strand (tripled ST + single gracilis) and the ALL graft, a single strand with the gracilis prolongation. ALL tibial tunnel will be performed with a 5mm drill, 1cm distal to the articular level, midway from the fibular head and Gerdy Tubercle, crossing the tibia toward its anteromedial cortex, 1cm distal to the ACL tunnel. Femoral ACL and ALL tunnels are coincident and located posterior and proximal to the lateral epicondyle. Intra-articular surgery will be performed in the same manner as comparative group. Gracilis prolongation is routed through the tibial ALL tunnel and then retrieved in the anteromedial aspect of the tibia, 1cm distal to the ACL tunnel entrance. ALL is fixed in full extension and neutral rotation, tying both graft extremities with 3 knots.
  Arms: Combined ACL and ALL

SUMMARY:
Persistent rotational instability after standard ACL reconstruction have been extensively described, and it has been shown to keep straight correlation with worse outcomes post-operatively (Chouliaras 2007, Kocher 2004). Anterolateral ligament (ALL) injury have been shown to play a relevant role in the genesis of rotational instability of the knee (Claes 2013, Helito 2013). Many anatomical publications have defined the ALL as a distinct ligament (Claes 2013). Meanwhile, some authors have proposed the association of ACL and ALL reconstruction in selected ACL-deficient individuals to further enhance knee stability postoperatively (Sonnery-Cottet 2015, Dodds 2014). Lack of consensus still predominates among ACL experts regarding the reliability of the combined ACL and ALL considering the controversy that involves both ALL anatomy and biomechanics (Guenther D 2016, Kittl C 2016). Clinical trials with high level of evidence and long term follow-up may be useful in order to determine the reliability of the combined procedure in the clinical setting.

So, the present study aims to compare the effectiveness of the combined ACL and ALL reconstruction with isolated ACL reconstruction in individuals with high-risk of ACL re-rupture, through a randomized controlled trial.

DETAILED DESCRIPTION:
Rotational knee stability is a topic with great interest among Anterior Cruciate Ligament (ACL) Reconstruction experts. Previous papers have questioned whether current ACL reconstruction techniques may provide adequate rotational stability in all ACL-deficient individuals, considering their broad spectrum of clinical presentations (Logan 2004, Ristanis 2005). Persistent rotational instability after standard ACL reconstruction have been extensively described, and it has been shown to keep straight correlation with worse outcomes post-operatively (Chouliaras 2007, Kocher 2004). Besides, lack of knee stability could lead to further chondral and meniscal lesions, which could enhance development of knee osteoarthritis (Stergiou 2007).

This discussion has gained increased attention after recent publications regarding the Anterolateral ligament (ALL), described as a structure whose lesion seems to worsen rotational instability when associated to ACL ruptures. (Claes 2013, Helito 2013, etc). Segond first described this ligament in 1897 as a "resistant fibrous band" located in the anterolateral knee compartment with a singular characteristic of tensioning in forced internal rotation (Segond 1879). Afterwards, some authors referred to this structure as a capsular thickening (Hughston 1976). More recently, various anatomical publications brought up this controversy, defining the ALL as a distinct ligament (Claes 2013, Dodds 2014, Helito 2015). Biomechanical data have shown straight correlation between its rupture and worsening of rotational stability, defined with a presence of an obvious positive pivot shift test (Claes 2013, Monaco 2012). Lack of consensus still exists regarding the validity of these findings, but many authors proposed the association of ACL and ALL reconstruction in selected ACL-deficient individuals, considering the theoretical biomechanical advantage of this procedure in promoting combined anteroposterior and rotational stability (Sonnery-Cottet 2015, Sonnery-Cottet 2017, Dodds 2014, Marcacci 2009). In a recent meta-analysis of randomized controlled trials, isolated ACL reconstruction techniques were compared to combined ACL and extra-articular reconstruction techniques and, although Lachman and pivot shift tests were superior in the combined ACL reconstruction group, functional scores were similar (Rezende 2015). Knee stiffness and infection, were also similar between groups, despite previous publications suggesting increased rates in the combined procedure (Anderson 2001, Sonnery-Cottet 2011). However, considering the lack of improvement of knee scores tests, the authors concluded it is still uncertain whether this increased stability surpasses the morbidity of adding an extra-articular procedure (Rezende 2015). In contrast to the obsolete extra-articular techniques included in the latter meta-analyses, anatomical ALL reconstruction techniques have been proposed to better replicate the anatomy of the anterolateral compartment (Sonnery-Cottet 2015). Promising results have been published in a recent prospective cohort study comparing combined ALL and ACL reconstruction with isolated ACL reconstruction techniques, using either hamstrings and bone-patellar-tendon bone grafts. Re-rupture rates were 3.1 times fold less in combined ACL and ALL procedure compared to isolated ACL with hamstrings and 2.3 times fold less compared to isolated ACL with bone-patellar-bone graft . The percutaneous ALL reconstruction technique described in this study not just reproduces more reliably the anatomy of the anterolateral compartment, but it is also less invasive diminishing the morbidity associated with the non-anatomic extra-articular reconstruction techniques, such as the iliotibial band tenodesis (Sonnery-Cottet 2017).

Many controversy still predominates among ACL experts not just regarding ALL in vitro studies, but also the debate about the reliability of the combined ACL and ALL procedure when bringing it to the clinical setting (Guenther D 2016, Kittl C 2016). Concerns have been raised about some aspects of the combined ACL and ALL procedure, in particular its theoretical potential in leading to an excessive knee constriction, as demonstrated in some biomechanical papers (Schon JM 2016). Experts opinions diverge about the potential long-term consequences of the combined ACL and ALL procedure; while defenders state that improved rotational instability should minimize degenerative consequences of a "sub-optimal" knee joint stability supposedly provided by an isolated intra-articular reconstruction, many other surgeons argue that knee osteoarthritis might the evolution of the abnormal kinematics of an overconstrained knee (Inderhaug E 2017, Schon JM 2016, Sonnery-Cottet B 2017). In order to resolve such lack of consensus, clinical trials with high level of evidence should be the priority in this field, with a long term follow-up, aiming to compare functional scores, knee stability tests and complications rates between isolated ACL and combined ACL and ALL reconstruction techniques.

So, the present study aims to compare the effectiveness of the combined ACL and ALL reconstruction with isolated ACL reconstruction in individuals with high risk of ACL re-rupture, through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 or 3 pivot shift test
* Chronic ACL lesions (>or= 1 year after lesion)

Exclusion Criteria:

* Previous knee surgeries
* Chondral grade IV knee lesions
* Concomitant knee ligament injuries, other than ACL and ALL ligaments
* Knee osteoarthritis
* Semitendinosus graft length shorter than 24mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
IKDC subjective part for functional outcome | 24 months
  International Knee Documentation Committee
Lysholm for functional outcome | 24 months
  Lysholm
KOOS for functional outcome | 24 months
  Knee injury and Osteoarthritis Outcome Score
Knee stability (subjective measures) | 24 months
  Lachman and pivot shift tests
Knee stability (objective measure) | 24 months
  Differential laxity (Rolimeter)

SECONDARY OUTCOMES:
Re-rupture | 24 months
  Presence of instability and pathological laxity postoperatively needing ACL revision (Middleton KK 2014).
Pain | 24 months
  Visual Analogue Scale (VAS)
Activity Level | 24 months
  Tegner

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Rezende, MD, Principal Investigator — research assistant
Locations (1):
- Federal University of Sao Paulo, Orthopedics and Traumatology Department (UNIFESP-EPM), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
No IPD plan established yet.

REFERENCES:
- [Background] Anderson AF, Snyder RB, Lipscomb AB Jr. Anterior cruciate ligament reconstruction. A prospective randomized study of three surgical methods. Am J Sports Med. 2001 May-Jun;29(3):272-9. doi: 10.1177/03635465010290030201. PMID 11394593
- [Background] Chouliaras V, Ristanis S, Moraiti C, Stergiou N, Georgoulis AD. Effectiveness of reconstruction of the anterior cruciate ligament with quadrupled hamstrings and bone-patellar tendon-bone autografts: an in vivo study comparing tibial internal-external rotation. Am J Sports Med. 2007 Feb;35(2):189-96. doi: 10.1177/0363546506296040. Epub 2007 Jan 23. PMID 17251174
- [Background] Claes S, Vereecke E, Maes M, Victor J, Verdonk P, Bellemans J. Anatomy of the anterolateral ligament of the knee. J Anat. 2013 Oct;223(4):321-8. doi: 10.1111/joa.12087. Epub 2013 Aug 1. PMID 23906341
- [Background] Dodds AL, Halewood C, Gupte CM, Williams A, Amis AA. The anterolateral ligament: Anatomy, length changes and association with the Segond fracture. Bone Joint J. 2014 Mar;96-B(3):325-31. doi: 10.1302/0301-620X.96B3.33033. PMID 24589786
- [Background] Guenther D, Rahnemai-Azar AA, Bell KM, Irarrazaval S, Fu FH, Musahl V, Debski RE. The Anterolateral Capsule of the Knee Behaves Like a Sheet of Fibrous Tissue. Am J Sports Med. 2017 Mar;45(4):849-855. doi: 10.1177/0363546516674477. Epub 2016 Dec 8. PMID 27932332
- [Background] Helito CP, Demange MK, Bonadio MB, Tirico LE, Gobbi RG, Pecora JR, Camanho GL. Anatomy and Histology of the Knee Anterolateral Ligament. Orthop J Sports Med. 2013 Dec 9;1(7):2325967113513546. doi: 10.1177/2325967113513546. eCollection 2013 Dec. PMID 26535259
- [Background] Hughston JC, Andrews JR, Cross MJ, Moschi A. Classification of knee ligament instabilities. Part II. The lateral compartment. J Bone Joint Surg Am. 1976 Mar;58(2):173-9. PMID 1254620
- [Background] Inderhaug E, Stephen JM, Williams A, Amis AA. Biomechanical Comparison of Anterolateral Procedures Combined With Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2017 Feb;45(2):347-354. doi: 10.1177/0363546516681555. Epub 2016 Dec 27. PMID 28027653
- [Background] Kittl C, El-Daou H, Athwal KK, Gupte CM, Weiler A, Williams A, Amis AA. The Role of the Anterolateral Structures and the ACL in Controlling Laxity of the Intact and ACL-Deficient Knee. Am J Sports Med. 2016 Feb;44(2):345-54. doi: 10.1177/0363546515614312. Epub 2015 Dec 10. PMID 26657572
- [Background] Kocher MS, Steadman JR, Briggs KK, Sterett WI, Hawkins RJ. Relationships between objective assessment of ligament stability and subjective assessment of symptoms and function after anterior cruciate ligament reconstruction. Am J Sports Med. 2004 Apr-May;32(3):629-34. doi: 10.1177/0363546503261722. PMID 15090377
- [Background] Logan MC, Williams A, Lavelle J, Gedroyc W, Freeman M. Tibiofemoral kinematics following successful anterior cruciate ligament reconstruction using dynamic multiple resonance imaging. Am J Sports Med. 2004 Jun;32(4):984-92. doi: 10.1177/0363546503261702. PMID 15150047
- [Background] Marcacci M, Zaffagnini S, Giordano G, Iacono F, Presti ML. Anterior cruciate ligament reconstruction associated with extra-articular tenodesis: A prospective clinical and radiographic evaluation with 10- to 13-year follow-up. Am J Sports Med. 2009 Apr;37(4):707-14. doi: 10.1177/0363546508328114. Epub 2009 Feb 3. PMID 19193599
- [Background] Monaco E, Ferretti A, Labianca L, Maestri B, Speranza A, Kelly MJ, D'Arrigo C. Navigated knee kinematics after cutting of the ACL and its secondary restraint. Knee Surg Sports Traumatol Arthrosc. 2012 May;20(5):870-7. doi: 10.1007/s00167-011-1640-8. Epub 2011 Aug 30. PMID 21877296
- [Background] Rezende FC, de Moraes VY, Martimbianco AL, Luzo MV, da Silveira Franciozi CE, Belloti JC. Does Combined Intra- and Extraarticular ACL Reconstruction Improve Function and Stability? A Meta-analysis. Clin Orthop Relat Res. 2015 Aug;473(8):2609-18. doi: 10.1007/s11999-015-4285-y. Epub 2015 Apr 7. PMID 25845949
- [Background] Ristanis S, Stergiou N, Patras K, Vasiliadis HS, Giakas G, Georgoulis AD. Excessive tibial rotation during high-demand activities is not restored by anterior cruciate ligament reconstruction. Arthroscopy. 2005 Nov;21(11):1323-9. doi: 10.1016/j.arthro.2005.08.032. PMID 16325082
- [Background] Schon JM, Moatshe G, Brady AW, Serra Cruz R, Chahla J, Dornan GJ, Turnbull TL, Engebretsen L, LaPrade RF. Anatomic Anterolateral Ligament Reconstruction of the Knee Leads to Overconstraint at Any Fixation Angle. Am J Sports Med. 2016 Oct;44(10):2546-2556. doi: 10.1177/0363546516652607. Epub 2016 Jul 12. PMID 27407088
- [Background] Sonnery-Cottet B, Archbold P, Zayni R, Bortolletto J, Thaunat M, Prost T, Padua VB, Chambat P. Prevalence of septic arthritis after anterior cruciate ligament reconstruction among professional athletes. Am J Sports Med. 2011 Nov;39(11):2371-6. doi: 10.1177/0363546511417567. Epub 2011 Aug 19. PMID 21856928
- [Background] Sonnery-Cottet B, Thaunat M, Freychet B, Pupim BH, Murphy CG, Claes S. Outcome of a Combined Anterior Cruciate Ligament and Anterolateral Ligament Reconstruction Technique With a Minimum 2-Year Follow-up. Am J Sports Med. 2015 Jul;43(7):1598-605. doi: 10.1177/0363546515571571. Epub 2015 Mar 4. PMID 25740835
- [Background] Sonnery-Cottet B, Barbosa NC, Vieira TD, Saithna A. Clinical outcomes of extra-articular tenodesis/anterolateral reconstruction in the ACL injured knee. Knee Surg Sports Traumatol Arthrosc. 2018 Feb;26(2):596-604. doi: 10.1007/s00167-017-4596-5. Epub 2017 Jun 12. PMID 28608009
- [Background] Stergiou N, Ristanis S, Moraiti C, Georgoulis AD. Tibial rotation in anterior cruciate ligament (ACL)-deficient and ACL-reconstructed knees: a theoretical proposition for the development of osteoarthritis. Sports Med. 2007;37(7):601-13. doi: 10.2165/00007256-200737070-00004. PMID 17595155